CLINICAL TRIAL: NCT06923436
Title: FROM THE INVISIBLE TO THE VISIBLE: Survey on the Psychological Well-being of Hospital Healthcare Workers
Brief Title: Survey of Psychological Well-being of Health Care Workers in the Hospital Setting
Acronym: IN-VISIBLE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7439
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Psychological Well Being; Stress Response; Professional Quality of Life; Resilience; Alexithymia; Spirituality; Coping Skills; Job-related Affective Well-being; Burnout, Healthcare Workers; Empathy Skills; Quality of Life Outcomes; Technostress
Keywords: Psychological well-being of health care workers in the hospital setting; work-related stress; emotional burden; Motivational aspects of health professionals; occupational well-being; Perceived Stress; Perceived stress from the intensive use of digital technology in work settings
MeSH Terms: conditions — Psychological Well-Being; Fractures, Stress; Affective Symptoms; Burnout, Psychological; Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital health workers: Hospital healthcare workers in departments most considered to be at risk of work-related stress (emergency, oncology)
  Interventions: Behavioral: Psychological Assessment

INTERVENTIONS:
Behavioral: Psychological Assessment — Collection of anamnestic and socio-demographic data, test administration repeated 4 months apart to monitor any changes

SUMMARY:
The psychological well-being of healthcare workers in hospital settings is a topic of growing interest in the scientific literature, given the crucial importance of their role in ensuring high-quality care. In addition, the Covid-19 pandemic health emergency has further accentuated the relevance of this issue, increasing anxiety and stress levels, testing the resilience and resistance of those working in care settings, revealing and highlighting how the accumulation of work-related stress can result in disabling pathologies for the caregiver, with an inevitable impact on the facility and care in general. Recent studies show that health care workers are particularly vulnerable to work-related stress, which can result from various factors such as high work demands, emotional pressure, irregular shifts, and interactions with critically ill patients. Burnout syndrome, characterized by emotional exhaustion, depersonalization and reduced personal accomplishment, is widely documented among hospital staff. Research indicates that burnout not only compromises the psychological health of healthcare workers, but also negatively affects the quality of care provided by increasing the risk of medical errors.

In light of these factors, it is crucial to deepen our understanding of the dynamics that influence psychological well-being and work-related stress in health care workers in order to develop effective interventions that can improve their quality of life and consequently the quality of care provided to patients.

Preliminary assessment of the emotional burden and motivational aspects of health care workers (showing what very often eludes a first glance, making visible something that is often invisible), along with effective stress management, would allow for greater ability to remain calm under pressure, reduced frustration, increased ability to make informed decisions, and to communicate effectively with patients and colleagues. These aspects translate into an image of a safer and more caring health care system in promoting better quality of care.

The aim of this project is to highlight the importance of psychological wellbeing for those working in health care settings and to promote attention to this area, also with a view to identifying possible interventions aimed at identifying preventive and protective factors in relation to health care workers.

The aim, therefore, is to show what is very often invisible at first sight, to make visible what is invisible: to explore, accommodate and contain areas of criticality and fragility in the context of work in health care settings, working on interventions aimed at the psychological well-being of workers.

DETAILED DESCRIPTION:
this work aims to recognise and legitimise the potential stressors of those who work in the health sector, with a focus on the most critical departments in terms of patient type and intervention, aware of the need to explore emotional experiences and professional needs from a prevention and protection perspective, in order to design effective interventions that promote the protection of operators' psychological well-being and strengthen their resilience factors. Drug-free, device-free, single-center, prospective longitudinal observational study with a total duration of 18 months.

Primary Objective: To record and describe over time some psychological dimensions related to the work activity of FPG workers, with a focus on contexts and departments considered more critical (for the type of activity or type of patients, such as the emergency area or oncology wards), in order to highlight possible areas of improvement and with respect to psychological well-being and Quality of Life (QoL) in the professional setting.

Secondary Objectives:

* Improving coping strategies, enhancing resilience, assessing aspects related to self-perception and self-efficacy in the work environment.
* Assess any correlations between what emerged from the psychological profile and: socio-demographic data, type of context in which one works, previous exposure to traumatic events, any psychological treatment.
* To assess how the motivation and/or over-involvement of operators in the relevant work contexts may be related to the development of work stress, which in turn could be a predictor with respect to issues inherent in the phenomena of absenteeism, work distress, job abandonment, transfer requests.

Sample size: 500 operators. Since this is an observational study whose analysis approach will be predominantly descriptive, no formal calculation of sample size based on hypothesis testing is planned. Based on the number of health care workers at the Fondazione Policlinico Gemelli IRCCS who meet the inclusion and exclusion criteria, we estimate that we can enroll approximately 500 subjects. As a general indication, this numerosity will allow us to estimate proportions with a maximum standard error of 0.022.

Methodology: Questionnaire administration at 2 times (T0 baseline, T1 after 4 months), with the possibility of questionnaire completion through the Microsoft Forms online platform.

All variables under study will be assessed in the first instance by descriptive statistical techniques. In detail, qualitative variables will be summarized through absolute frequencies and percentages. As for the quantitative variables, their distribution will first be assessed using the Shapiro Wilk test, then where normally distributed they will be expressed as mean and standard deviation (SD), otherwise as median and interquartile range (IQR).

The primary endpoint related to the domain of psychological and occupational well-being, which is purely exploratory, will therefore be analyzed in terms of descriptive statistics, as reported above. The same approach will be followed for the assessment of the domains of relational and occupational well-being, coping strategies, and behavioral All questionnaires will be analyzed with reference to each individual scale, both in terms of overall score and with respect to individual items and through correlation with other tests. Changes between T0 and T1 will be investigated using paired data tests with parametric or nonparametric approach depending on the distribution of the variables themselves. Graphical representations will also be used to better interpret and communicate the results. Data analysis will be conducted using IBM-SPSS v.28.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Work activity carried out in departments classified as at risk for work-related stress (emergency care, oncology...)
* Willingness to participate in the study and the ability to understand and sign the informed consent form.

Exclusion Criteria:

* Psychological/psychiatric comorbidities
* Inability to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare workers, with a focus on contexts and departments considered more critical (due to the type of activity or the type of patients, such as the emergency area or oncology departments).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of indicators of work-related psychological well-being using the Maslach Scale (MBI), with evaluation of any differences between a Baseline, and after 4 months | From enrollment (Time 0) to 4 weeks (Time 1)
  The Maslach Burnout Inventory (MBI) is a widely used psychological assessment instrument developed for measuring and evaluating burnout of individuals in various professional settings. The MBI is a self-report questionnaire whose purpose is to measure the various dimensions of burnout that include emotional exhaustion, depersonalization and reduced personal accomplishment.
  Consisting of 22 items, each of which includes 6 different response grades on a Likert scale, this test facilitates the creation of tailored interventions and strategies to prevent or address burnout effectively.
Assessment of indicators of work-related Stress, using the Perceived Stress Scale (PSS), with evaluation of any differences between a Baseline, and after 4 months. | From enrollment (Time 0) to 4 weeks (Time 1)
  Perceived Stress Scale (PSS) is the most widely used instrument for assessing perceived stress in individuals aimed at measuring the degree to which situations in one's life are rated as stressful.
  It is a test consisting of 10 questions in which the individual's feelings and thoughts over the previous month are investigated and asked to express the frequency with which these occur using a Likert scale of 5 different grades. Minimum score is 0, maximum score is 40.
  The items were developed so that they can detect how unpredictable, uncontrollable and overloaded individuals feel their lives are.
  Scores from 0 to 13: low perceived stress Scores from 14 to 26: moderate perceived stress Scores froom 27 to 40: high perceived stress

SECONDARY OUTCOMES:
Assessment of coping styles through the Brief-COPE questionnaire, with evaluation of any differences between a Baseline, and after 4 months. | From enrollment (Time 0) to 4 weeks (Time 1)
  The Brief-COPE questionnaire is a self-report questionnaire consisting of 25 items. The questionnaire asks to assess how often the subject enacts--in difficult or stressful situations--that particular coping process; there are four response options, from "I usually don't" to "I almost always do." Fifteen different coping mechanisms are considered: Activity, Planning, Suppression of competitive activities, Containment, Seeking information, Seeking understanding, Emotional outburst, Positive reinterpretation and growth, Acceptance, Devotion to religion, Humor, Denial, Behavioral detachment, Mental detachment, Drug or alcohol use.
Evaluation of motivation/attachment to one's work through the Job-related Affective Well-being Scale (JAWS), with evaluation of any differences between a Baseline, and after 4 months. | From enrollment (Time 0) to 4 weeks (Time 1)
  The Job-related Affective Well-being Scale (JAWS) is a 30-item scale designed to assess individuals' emotional reactions to their work.
  Each item represents an emotion, and respondents are asked how often they have experienced each one at work over the past 30 days. Responses are given on a five-point scale corresponding to the options: Never, Rarely, Sometimes, Quite often, Extremely often, or Always.
  The JAWS encompasses a wide range of emotional experiences, both negative and positive. The emotions can be categorized into four subscales, structured along two dimensions: pleasantness and arousal (intensity).
Evaluation of Empathy with the Balanced Emotional Empathy Scale - BEES, with evaluation of any differences between a Baseline, and after 4 months. | From enrollment (Time 0) to 4 weeks (Time 1)
  The Balanced Emotional Empathy Scale (BEES) is a self-report questionnaire designed to measure the level of empathy.
  It consists of 30 items with both positive and negative connotations. The statements in the scale refer to real-life situations, and agreement is expressed using a 9-point Likert scale.
  The total score, calculated based on all responses to the various statements, can range from a maximum of 3 to a minimum of -3. A score of 0±0.5 corresponds to an average level of empathy. Positive values above 0 indicate above-average empathy, with higher values representing greater empathy, while negative values below 0 indicate below-average empathy.
Assessment of Quality of Life in the Professional Context through the Professional Quality of Life Scale (ProQOL), with evaluation of any differences between a Baseline, and after 4 months. | From enrollment (Time 0) to 4 weeks (Time 1)
  A 30-item questionnaire designed to measure compassion fatigue, job satisfaction, and burnout among healthcare professionals. It is useful for workers engaged in emotional labor and professionals exposed to traumatic situations. Professional Quality of Life refers to the quality one experiences in relation to their work as a helper. Both the positive and negative aspects of performing one's job influence professional quality of life.
  The ProQOL measures three aspects of professional quality of life: Compassion Satisfaction (the pleasure derived from being able to do one's job well); Burnout (exhaustion, frustration, anger, and depression related to work); Secondary Traumatic Stress (experiencing fear in relation to primary or secondary work-related trauma).
Assessment of Spiritual Well-being (by FACIT-Sp-12), with evaluation of any differences between a Baseline, and after 4 months. | From enrollment (Time 0) to 4 weeks (Time 1)
  FACIT-Sp-12 (The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being) is a test designed to measure spiritual well-being. It consists of 12 items, evaluated on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). When completing the questionnaire, respondents are asked to refer to the past 7 days. There are 2 reverse-scored items (Sp4 and Sp8). The scale is primarily divided into three dimensions: meaning in life, sense of peace, and faith. To obtain the total score, the values from these three domains are summed. There are no cut-off scores: the higher the score, the better the individual's spiritual well-being
Evaluation of technostress in workplace settings, with evaluation of any differences between a Baseline, and after 4 months. | From enrollment (Time 0) to 4 weeks (Time 1)
  The Technostress Creators Scale (TCS) measures how various aspects of technology can lead to discomfort, anxiety, and dissatisfaction among employees. It identifies five key factors, known as "technostress creators," that affect workers' psychological well-being:
  Overload (excessive technological demands), Invasion (technology intruding into personal life), Complexity (difficulty in understanding and using technology), Uncertainty (constant changes in technology), and Insecurity (fear of job loss due to technological advancements).
  The goal of the TCS is to help organizations to create more balanced and sustainable work environments. This can be achieved through targeted interventions such as training support, redefining digital processes (Min tot score: 11; Max tot score: 55)
  Subscale Scores:
  Techno-overload: from 4 to 20 Techno-invasion: from 3 to 15 Techno-complexity: from 4 to 20 Higher scores indicate a greater level of perceived technostress within each respective dimension.
Assessing Resilience (with RS-14) with evaluation of any differences between a Baseline, and after 4 months. | From enrollment (Time 0) to 4 weeks (Time 1)
  The scale consists of 14 items, each rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree).
  All items have a positive score, with a minimum possible score of 14 and a maximum of 98.
  The scoring interpretation is as follows:
  <56 indicates a very low level of resilience, 57-64 indicates a low level of resilience, 65-73 indicates a moderately low level of resilience, 74-81 indicates a moderate level of resilience, 82-90 indicates a moderately high level of resilience, >91 indicates a high level of resilience.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Callegari C, Bertu L, Lucano M, Ielmini M, Braggio E, Vender S. Reliability and validity of the Italian version of the 14-item Resilience Scale. Psychol Res Behav Manag. 2016 Oct 3;9:277-284. doi: 10.2147/PRBM.S115657. eCollection 2016. PMID 27757055
- [Background] Palmieri G, Evans C, Hansen V, Brancaleoni G, Ferrari S, Porcelli P, Reitano F, Rigatelli M. Validation of the Italian version of the Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM). Clin Psychol Psychother. 2009 Sep-Oct;16(5):444-9. doi: 10.1002/cpp.646. PMID 19701881
- [Background] Maresca G, Corallo F, Catanese G, Formica C, Lo Buono V. Coping Strategies of Healthcare Professionals with Burnout Syndrome: A Systematic Review. Medicina (Kaunas). 2022 Feb 21;58(2):327. doi: 10.3390/medicina58020327. PMID 35208650
- [Background] Pollock A, Campbell P, Cheyne J, Cowie J, Davis B, McCallum J, McGill K, Elders A, Hagen S, McClurg D, Torrens C, Maxwell M. Interventions to support the resilience and mental health of frontline health and social care professionals during and after a disease outbreak, epidemic or pandemic: a mixed methods systematic review. Cochrane Database Syst Rev. 2020 Nov 5;11(11):CD013779. doi: 10.1002/14651858.CD013779. PMID 33150970
- [Background] Laserna Jimenez C, Casado Montanes I, Carol M, Guix-Comellas EM, Fabrellas N. Quality of professional life of primary healthcare nurses: A systematic review. J Clin Nurs. 2022 May;31(9-10):1097-1112. doi: 10.1111/jocn.16015. Epub 2021 Aug 27. PMID 34453386
- [Background] National Academies of Sciences, Engineering, and Medicine; National Academy of Medicine; Committee on the Future of Nursing 2020-2030; Flaubert JL, Le Menestrel S, Williams DR, Wakefield MK, editors. The Future of Nursing 2020-2030: Charting a Path to Achieve Health Equity. Washington (DC): National Academies Press (US); 2021 May 11. Available from http://www.ncbi.nlm.nih.gov/books/NBK573914/ PMID 34524769
- [Background] Trumello C, Bramanti SM, Ballarotto G, Candelori C, Cerniglia L, Cimino S, Crudele M, Lombardi L, Pignataro S, Viceconti ML, Babore A. Psychological Adjustment of Healthcare Workers in Italy during the COVID-19 Pandemic: Differences in Stress, Anxiety, Depression, Burnout, Secondary Trauma, and Compassion Satisfaction between Frontline and Non-Frontline Professionals. Int J Environ Res Public Health. 2020 Nov 12;17(22):8358. doi: 10.3390/ijerph17228358. PMID 33198084